CLINICAL TRIAL: NCT07217938
Title: TRADstat: Novel Treatment of Radiation Associated Dysphagia With Statins
Brief Title: Novel Treatment of Radiation Associated Dysphagia With Statins
Acronym: TRADstat
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121555
Record Dates: First submitted 2025-09-09; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Radiation-associated Dysphagia; Head &Amp; Neck Cancer
Keywords: Radiation-associated dysphagia; Dysphagia; Head & neck cancer; Pravastatin
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders | interventions — Pravastatin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study (Experimental): Single arm study
  Interventions: Drug: Pravastatin 40 Mg Oral Tablet

INTERVENTIONS:
Drug: Pravastatin 40 Mg Oral Tablet — This trial will incorporate Pravastatin 40 mg as an off-label use for the treatment of radiation-associated dysphagia.

SUMMARY:
The aim of this trial is to examine the feasibility, acceptability, and potential efficacy of a 12-month course of pravastatin as an antifibrotic agent for managing dysphagia (swallowing problems) in patients previously treated with radiotherapy for head and neck cancer (HNC). The purpose is to assess whether pravastatin, a medication approved in Australia for cholesterol management, can improve swallowing in people with long-term radiation-associated dysphagia following HNC treatment.

The trial will recruit 48 patients, with an anticipated accrual period of approximately 6 months. Eligible patients will be identified from the Principal Investigator's current study, ERADICATE, or through referral by a radiation oncologist or speech pathologist diagnosing radiation-induced dysphagia.

Participants will receive 40 mg of pravastatin daily for up to 12 months, with swallowing assessments conducted before, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent using the TRADstat PICF
2. Patients aged 18 years or older at screening
3. Received curative intent (chemo)radiotherapy to the nasopharynx, oropharynx, hypopharynx or larynx at least 2 years prior to screening
4. Moderate-severe RAD using validated cut-offs (PAS score > 3 and/or DIGEST grading ≥ 2), identified on a VFSS conducted within the last 12 months
5. Adequate kidney function defined as estimated glomerular filtration rate (eGFR) ≥ 40 ml/min
6. Adequate hepatic function defined as:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than 2 times the upper normal limit (ULN)
   * Bilirubin level at least 1.5 times lower than the ULN
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2 (Appendix 1)

Exclusion Criteria:

1. Known hypersensitivity to pravastatin and/or any excipients
2. Diagnosis of myasthenia (muscle weakness)
3. History of head or neck surgery, other than excisional biopsy or post treatment neck dissection
4. Known active malignancy
5. Currently taking statin medication
6. Currently taking prohibited medicines (long-term steroids or drugs listed under Section 8.4)
7. History of severe heart failure; a history of muscle toxicity during previous treatments with fibrates or statins; a history of hereditary muscle diseases
8. Known medical condition(s) that may impact swallowing function (e.g., stroke, neurological conditions, tracheostomy)
9. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the pravastatin to treat radiation-associated dysphagia | From enrolment to the end of 12 months of pravastatin use
  A Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) grade decrease of at least 1-point after 12 months of pravastatin from registration. The DIGEST scale ranges between 0 to 4, with 4 being the worst outcome.
Feasibility of the use of pravastatin to treat radiation-associated dysphagia | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Percentage of eligible patients who consent to recruitment and percentage of recruited (registered) patients who remain on pravastatin for 12 months and complete the 6-month follow-up assessment

SECONDARY OUTCOMES:
Acceptability of trial methods and procedures and acceptability of pravastatin | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Acceptability of trial methods and procedures, and acceptability of pravastatin: Theoretical Framework of Acceptability (TFA) questionnaire total score. The TFA used in this study ranges between 11 - 55 and higher scores represent better acceptability.
Tolerability of pravastatin | From the start of pravastatin therapy until the completion of 12 months of therapy
  Tolerability of pravastatin: percentage of patients who cease pravastatin (patient or clinician choice) due to pravastatin related toxicity using Common Toxicity Criteria for Adverse Events, Version 5.0 (CTCAE v5.0), and the range is 0 to 5, with 5 being the worst outcome
Safety of pravastatin use | From the start of pravastatin therapy until the completion of 12 months of therapy
  Safety of pravastatin use: percentage of patients who experience ≥ Grade 2 toxicity (as per Common Toxicity Criteria for Adverse Events, Version 5.0 [CTCAE v5.0], and the range is 0 to 5, with 5 being the worst outcome)
Immune-biomarker outcome | At baseline and after 12 months of pravastatin treatment.
  Immune-biomarker outcome: collection of 10 mL edta tube for the immune-biomarker analysis. Specific biomarker selection still under process.

OTHER OUTCOMES:
Clinician-rated penetration/aspiration | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Clinician-rated penetration/aspiration: Penetration-Aspiration scale (PAS) score assessed via videofluoroscopy swallow studies (VFSS), the range is 1 to 8, with 8 representing the worst outcome.
Biomechanical swallowing measures | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Bio-mechanical swallowing measures: using the Computational Analysis of Swallowing Mechanics (CASM) via VFSS, no specific range is available, however ; higher values represent better outcome.
Clinician-rated functional status | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Clinician-rated functional status: Performance Status Scale for Head and Neck Cancer Patients (PSS-HN) subscale scores, the range is between 0 to 100, with higher values representing better outcomes.
Trismus (limitations in mouth opening) | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Trismus (limitations in mouth opening): Maximal-interincisal opening as measured using the TheraBite® Range-of-Motion scale, the range is between 0 to 70 mm, with higher values representing better outcomes.
Patient-reported swallowing problem severity | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Patient-reported swallowing problem severity: Eating Assessment Tool (EAT-10) total score, the range is between 0 to 40, with higher values representing worse outcomes.
Patient-reported swallowing-related QoL: | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Patient-reported swallowing-related QoL: M.D. Anderson Dysphagia Inventory (MDADI) global score, the range is between 20 to 100, with higher values representing better outcomes.
Patient-reported lymphoedema and fibrosis symptoms and impacts | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Patient-reported lymphoedema and fibrosis symptoms and impacts: Head and Neck Lymphedema and Fibrosis Symptom Inventory (HN-LEF), the range is between 0 to 165, with higher values representing worse outcomes.
Nutritional outcomes | From the start of pravastatin therapy to 6 months of follow up after the completion of 12 months of pravastatin therapy (total estimated time duration 18 months)
  Nutritional outcomes: Weight and feeding tube use (percentage of nutritional requirements taken via gastrostomy tube versus oral intake)

IPD SHARING:
Plan to Share IPD: No
Date will not be shared due to ethical reasons.

REFERENCES:
- [Background] Bourgier C, Auperin A, Rivera S, Boisselier P, Petit B, Lang P, Lassau N, Taourel P, Tetreau R, Azria D, Bourhis J, Deutsch E, Vozenin MC. Pravastatin Reverses Established Radiation-Induced Cutaneous and Subcutaneous Fibrosis in Patients With Head and Neck Cancer: Results of the Biology-Driven Phase 2 Clinical Trial Pravacur. Int J Radiat Oncol Biol Phys. 2019 Jun 1;104(2):365-373. doi: 10.1016/j.ijrobp.2019.02.024. Epub 2019 Feb 15. PMID 30776452